CLINICAL TRIAL: NCT02232828
Title: Selective or Stepwise Removal of Deep Caries in Deciduous Molars: A Multi-center Randomized Controlled Trial
Brief Title: Selective or Stepwise Removal of Deep Caries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Rheinisch-Westfälische Technische Hochschule RWTH Aachen, Germany (Unknown); University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Falk Schwendicke, OA Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARIEX2or1
Record Dates: First submitted 2014-08-29; First posted 2014-09-05 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Selective removal (Experimental)
  Interventions: Procedure: Selective removal
- Stepwise removal (Active Comparator)
  Interventions: Procedure: Stepwise removal

INTERVENTIONS:
Procedure: Selective removal — Caries removal in the periphery including the enamel-dentinal junction will be performed using rose head burs and/or an excavator until hard, dry dentin remains. Pulpo-proximal caries will be removed until leathery, slightly moist and reasonably soft dentin remains. Operating dentists will be calibrated prior to study commencement regarding these criteria using extracted teeth. Moisture control will be performed using cotton rolls and continuous aspiration. Restoration will be performed adhesively, with a self-etching one-bottle adhesive (G-aenial bond, GC, Bad Homburg, Germany) and a compomer material (Dyract, Dentsply Detray, Konstanz, Germany) being used.
  Arms: Selective removal
Procedure: Stepwise removal — Caries removal in the periphery including the enamel-dentinal junction will be performed using rose head burs and/or an excavator until hard, dry dentin remains. Pulpo-proximal caries will be removed until leathery, slightly moist and reasonably soft dentin remains. Operating dentists will be calibrated prior to study commencement regarding these criteria using extracted teeth. Moisture control will be performed using cotton rolls and continuous aspiration. Restoration will be performed adhesively, with a self-etching one-bottle adhesive (G-aenial bond, GC, Bad Homburg, Germany) and a compomer material (Dyract, Dentsply Detray, Konstanz, Germany) being used.
  If allocated to stepwise excavation, the second excavation will now be performed as described until only hard, dry dentin remains. Restoration will again be provided adhesively as described.
  Arms: Stepwise removal

SUMMARY:
Background: For treating deep caries lesions, selective or stepwise, i. e. one- and two-step incomplete excavation seems advantageous compared with complete caries removal. However, current evidence regarding the success, as defined by not requiring any re-treatments, or survival of teeth after different excavations is insufficient for definitive recommendation, especially when treating deciduous teeth. Moreover, restoration integrity has not been comparatively analyzed longitudinally, and neither patients', dentists' or parents' preferences nor the clinical long-term costs emanating from both initial and re-treatments have been reported yet.

Our primary hypothesis is that success rates differ significantly between selectively and stepwise excavated teeth. Secondary hypotheses are that restoration integrity is assumed to significantly differ between selectively and stepwise excavated teeth.

DETAILED DESCRIPTION:
The treatment of deep caries lesions is associated with significant risks for the pulp, including pulpal exposure and post-operative pulpal complications, which might eventually compromise the retention of the tooth [1]. Moreover, treating deep lesions might be associated with pain and subjective burden both during and after treatment and might generate long-term costs due to re-treatments being required [2, 3].

For deciduous teeth, various treatments for deep lesions have been described: Complete excavation aims at removing all infected and affected carious dentin, with the inherent risk of pulpal exposure. In contrast, stepwise, i. e. two-step excavation leaves carious dentin after the initial excavation step, then seals residual caries under a temporary restoration, and re-enters the cavity in a second step to eventually attempt complete excavation. This approach is thought to facilitate arrest and remineralization of the lesion and to induce development of tertiary dentin, thereby reducing the risk of pulpal exposure and post-operative complications after the second excavation step [4, 5]. Since several studies found sealed residual lesions to be clinically and microbiologically arrested, the need to re-enter was increasingly questioned within the last decade [6]. Selective, i. e. one-step incomplete or partial excavation seals carious dentin under a definitive restoration, omitting any re-entry [7]. Sealing the lesion is thought to deprive residual bacteria from dietary carbohydrates and was found to exert significant antibacterial effects, thus arresting the lesion [8, 9].

However, doubts remain regarding the effects of sealed carious dentin on the long-term quality of the restoration [10]. Moreover, it remains unknown if patients prefer one of both treatments, which might be especially relevant when treating children. Several studies comparing complete with selective or stepwise excavation of deciduous teeth have been published, but only one three-arm study compared selective with stepwise excavation of primary teeth (Tab. 1). In addition, none of these studies assessed patient- or dentists-centered outcomes, i. e. preferences, or analyzed clinically assessed long-term costs emanating from both excavations.

Objectives and Hypotheses The study aims at comparing the success, i. e. the probability of not requiring any re-interventions, and the survival, i. e. the probability of not requiring tooth removal, of selectively versus stepwise excavated vital, non-symptomatic deciduous molars with deep lesions. In addition, we assess the restoration integrity of selectively versus stepwise excavated deciduous molars, evaluate the preference of patients, parents and dentists for one of both strategies, and comparatively assess the costs associated with each strategy.

Our primary hypothesis is that success rates differ significantly between selectively and stepwise excavated teeth. Secondary hypotheses are that restoration integrity is assumed to significantly differ between selectively and stepwise excavated teeth. Moreover, we hypothesize that patients', parents' and dentists' preference is significantly different for selective versus stepwise excavated teeth. Eventually, both initial and long-term costs of excavation methods are supposed to significantly differ.

The planned study is a secondary care-based prospective, multi-center two-arm, parallel-group, randomized controlled trial at three pediatric university dental clinics in Germany. We plan to enroll 300 patients with one or more deeply carious, sensitive and non-symptomatic deciduous molar. One molar per patient will be randomly allocated to receive one of two treatments (selective or stepwise excavation). Total follow-up time will be three years after completion of the initial treatment. Success, survival and restoration integrity will be assessed after one, two and three years. Patients', parents' and dentists' preference will be assessed after each treatment using visual-analogue scale or Likert-rating scales. Costs will be assessed for initial and follow-up treatments and will be based on a micro-costing approach.

ELIGIBILITY:
Inclusion Criteria:

* Children 3-9 yr
* Good general health
* Minimum one active deep (D3) occlusal/occlusal-proximal, one-/two-surface caries lesion

Exclusion Criteria:

* Participating in other study
* Plan to move or not resident
* Systemic disease or general disability
* Expected limited compliance
* Known allergy to study material expected exfoliation within 18 month

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Success (re-intervention required no/yes) | 36 month
  The primary outcome of the study will be success (i. e. not requiring any re-intervention).

SECONDARY OUTCOMES:
Survival (tooth removal required no/yes) | 36 months
  Secondary outcomes will include survival (i. e. not requiring extraction).
Restoration integrity (scored as alpha, beta, gamma, delta) | 36 months
  Restoration integrity will be assessed via modified USPHS-criteria.
Patients' subjective assessment of the treatment (0-10) | 0 months (directly after treatment)
  Patients' subjective assessment of the treatment will be recorded using visual-analogue scale. For stepwise excavation, assessments will be performed twice and mean VAS-results calculated.
Dentists' subjective assessment (1-6) | 0 months (directly after treatment)
  Dentists' subjective assessment of the treatment will be reported using grades from 1 (very good) to 6 (very bad).
Parents' subjective assessment (1-6) | 0 months (directly after treatment)
  similar to dentists' assessment
Treatment costs (Euro) | 36 months
  Total treatment costs (calculated by combining costs for staff, as assessed by time required for the procedures and the number of personnel involved, and costs for transportation of patients or materials) for both initial and follow-up treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Falk Schwendicke, OA Dr., Principal Investigator — Chatrite Berlin, Germany; Sebastian Paris, Prof. Dr., Study Chair — Charite Berlin, Germany; Christian Finke, OA Dr., Principal Investigator — Charite Berlin, Germany; Marina A. Petrou, Dr., Principal Investigator — Uniklinic RWTH Aachen, Germany; Christian Spleith, Prof. Dr., Principal Investigator — University Greifswald, Germany; Ruth Santamaria, Dr., Principal Investigator — University Greifswald, Germany
Locations (4):
- Germany (4):
  - Ernst-Moritz-Arndt University of Greifswald, Präventive Zahnmedizin und Kinderzahnheilkunde, Greifswald, Mecklenburg-Vorpommern
  - Uniklinik RWTH Aachen; Klinik für Zahnerhaltung, Parodontologie und Präventive Zahnheilkunde, Aachen, North Rhine-Westphalia
  - CharitéCentrum für Zahn-, Mund- und Kieferheilkunde der Charité - Universitätsmedizin Berlin, Abteilung für Kieferorthopädie, Orthodontie und Kinderzahnmedizin, Berlin, State of Berlin
  - CharitéCentrum für Zahn-, Mund- und Kieferheilkunde der Charité - Universitätsmedizin Berlin; Abteilungen für Zahnerhaltung und Präventive Zahnheilkunde, Berlin, State of Berlin

REFERENCES:
- [Derived] Elhennawy K, Finke C, Paris S, Reda S, Jost-Brinkmann PG, Schwendicke F. Selective vs stepwise removal of deep carious lesions in primary molars: 24 months follow-up from a randomized controlled trial. Clin Oral Investig. 2021 Feb;25(2):645-652. doi: 10.1007/s00784-020-03536-6. Epub 2020 Aug 28. PMID 32857210
- [Derived] Elhennawy K, Finke C, Paris S, Reda S, Jost-Brinkmann PG, Schwendicke F. Selective vs stepwise removal of deep carious lesions in primary molars: 12-Months results of a randomized controlled pilot trial. J Dent. 2018 Oct;77:72-77. doi: 10.1016/j.jdent.2018.07.011. Epub 2018 Jul 17. PMID 30025748
- [Derived] Schwendicke F, Schweigel H, Petrou MA, Santamaria R, Hopfenmuller W, Finke C, Paris S. Selective or stepwise removal of deep caries in deciduous molars: study protocol for a randomized controlled trial. Trials. 2015 Jan 6;16:11. doi: 10.1186/s13063-014-0525-9. PMID 25560779